CLINICAL TRIAL: NCT06050486
Title: A Mentalization-based Treatment for Children (MBT-C) of Parent(s) With Borderline Personality Disorder: A Pilot Study
Brief Title: A Mentalization-based Intervention for Children of Parent(s) With Borderline Personality Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minho (Other)
Responsible Party: Principal Investigator, Bárbara Figueiredo, Associate Professor with Aggregation, University of Minho
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEICSH 062/2021; 2020.08588.BD (Other Grant/Funding Number: Foundation for Science and Technology (FCT))
Record Dates: First submitted 2023-09-15; First posted 2023-09-22 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Child's Internalizing and Externalizing Problems
MeSH Terms: interventions — Mentalization-Based Therapy

STUDY DESIGN:
Intervention Model Description: The interventional model is a simple one-arm study (intervention), with 3 assessment waves (pretest, posttest and follow-up).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1: Intervention (Experimental): Participants in Arm 1 receive a psychological intervention (MBT-C).
  Interventions: Behavioral: Mentalization-based treatment for children (MBT-C)

INTERVENTIONS:
Behavioral: Mentalization-based treatment for children (MBT-C) — MBT-C is a time-limited intervention designed to resolve the child's emotional or behavioral problems and to promote resilience, by promoting the child's and parent's mentalizing capacities. It is composed by 1) an assessment phase, composed of 3 to 4 sessions, with the family, the child and the parent(s), 2) an intervention phase, composed of a minimum block of 12 individual sessions with the child and parallel sessions for the parent(s), that can be repeated up to three times (i.e., maximum of 36 sessions), and 3) a booster session 3 to 12 months after the last session. In this clinical trial, MBT-C will be composed of: 3 assessment sessions; 12 individual sessions with the child, plus 6 parallel individual sessions with the parent with BPD; 1 booster family session, 3 months after the last session.

SUMMARY:
Background and study aims? Parents with borderline personality disorder (BPD) can present parenting difficulties such as expressions of hostility, low sensitivity, and overprotection. These parenting problems are associated with adverse outcomes for the offspring, namely, borderline features, depression, internalizing and externalizing problems, and interpersonal difficulties. Intervention studies with parent(s) who have borderline personality disorder show promising results regarding the improvement of parenting skills and parent-infant relationship. However, very few assess their effect on child's mental health and development. This study aims to evaluate the acceptability, feasibility and preliminary effectiveness of a mentalization-based clinical intervention, directed to school-aged children of mothers and/or fathers with borderline personality disorder, to reduce child mental health problems, in the short- and medium-term.

Who can participate? School-aged children (5 to 12 years of age), with mental health problems (CBCL internalizing and/or externalizing scores must be T = 60 or above), and their mothers and/or fathers (> 18 years of age) with subclinical or clinical BPD.

What does the study involve? Mother and/or father with BPD complete an online survey and an online interview. If available, the other parent and the child's teacher complete an online survey, separately. The child completes an online task with a researcher's assistance. After, participants are assigned to an intervention group (one arm, pre-posttest study). Participants receive a mentalization-based treatment for children (MBT-C), starting one week after the pre-test. MBT-C is a psychological intervention designed to resolve the child's mental health problems and promote resilience by promoting the child's and parent's mentalizing capacities. It aims to be delivered by a mental healthcare professional trained in MBT-C. In this clinical trial MBT-C will be composed of: 3 assessment sessions; 12 individual sessions with the child, plus 6 parallel individual sessions with the parent with BPD; 1 follow-up family session, 3 months after the last session. Assessment sessions are composed of one family session, one session with the child and one session with the parent. Sessions with child are in-site and sessions with parent can be on-line or in-site, according to the parents' preference. Sessions have a weekly frequency and a 50-60 minutes duration each. One week after the last intervention session participants repeat the same assessments completed before MBT-C. In addition, child and mother and/or father with BPD complete separately an online satisfaction survey and an online interview to assess participants experiences with MBT-C.

The investigators expect that after receiving MBT-C the child's mental health problems will have significantly decreased and to obtain information on the feasibility of a future large-scale clinical trial and retrospective acceptability of MBT-C with this specific population.

What are the possible benefits and risks of participating? This intervention aims to resolve child's mentals mental health problems. Patients who do not meet the inclusion criteria to participate, do not consent, or withdraw from the trial will be offered a debrief and the possibility of being referred to individualized psychological support or other if needed. If child's mental health problems are not resolve by the end of MBT-C the same possibility will be offered. At the end of MBT-C mother and/or father with BPD will be referred to individual therapy, if needed and not already receiving. Intervention with BPD parents can present challenges, such as ambivalence within the therapeutic relationship (high idealization versus therapist rejection), and high drop-out rates. To overcome these difficulties, the therapist should be knowledgeable about BPD, foster a secure-based relationship with the parent and child, and maintain an empathetic stance. It is possible for parent(s) with BPD to maltreat or abuse their children, in which case child protective services must be contacted and informed. The same procedure must be adopted in case of substantial substance abuse.

ELIGIBILITY:
Inclusion Criteria Child:

* have a mother and/or father with subclinical or clinical symptoms of BPD;
* present internalizing and/or externalizing problems (i.e., ≥60 in the internalizing and/or externalizing scale of CBCL 6-18);
* be 5-12 years old.

Inclusion Criteria Parent(s):

* have subclinical or clinical symptoms of BPD;
* have a school-aged child (5-12 years of age) with internalizing and/or externalizing problems.

Exclusion Criteria Child:

* unable to read/speak Portuguese;
* comorbidity with a neurodevelopmental disorder (i.e., autism spectrum disorder with moderate to severe impairment; moderate to severe cognitive deficit);
* doesn´t live partially or fully with parent with BPD;
* already receiving psychological counselling.

Exclusion Criteria Parent(s):

* unable to read/speak Portuguese;
* comorbidity with another mental health disorder that could interfere with intervention viability (i.e., schizophrenia spectrum or other psychotic disorders; substance-related and addictive disorders, except caffeine, tobacco and cannabis).

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Child Behavior Checklist | Child is assessed with CBCL at 3 time-points: pretest (one to two weeks before the first session); posttest (one week after the last session); follow-up (3 months after the last session).
  CBCL is a parent reported questionnaire composed of 113 items that seek to assess behavioral and emotional problems in children from 1.5 to 18 years of age. It is a component of the Achenbach System (ASEBA). The items are scored on a 3-point scale (0 = "Not true (as far as we know)", 1 = "Somewhat or sometimes true" and "2 = very true or often true"). It comprises three scales: (1) Internalizing problems; (2) Externalizing problems; (3) Total Score. The cutoff point of the questionnaire is T Score = 60 or more, on all three scale, indicating a clinical level of the child's emotional and behavioral problems.

SECONDARY OUTCOMES:
Structured Clinical Interview for DSM-IV Axis II Personality Disorders | Parent is assessed at 3 time-points: pretest (one to two weeks before the first session); posttest (one week after the last session); follow-up (3 months after the last session).
  SCID-II is a semistructured diagnostic interview that assesses 10 Axis II personality disorders from the Diagnostic and Statistical Manual of Mental Disorders, 4th Ed (DSM-IV; APA, 2000), and the depressive and passive-aggressive personality disorders (included in DSM-IV's appendix). It can be used to diagnose Axis II disorders categorically (present or absent) and dimensionally (according to the number of criteria met for each diagnosis).
Emotional regulation checklist | Child is assessed at 3 time-points: pretest (one to two weeks before the first session); posttest (one week after the last session); follow-up (3 months after the last session).
  ERC is a parent or teacher reported questionnaire composed of 24 items to assess emotion regulation competencies in children from 6 to 12 years of age. The items are measured on a 4-point Likert scale (1 = never; 4 = almost always), with two subscales: emotion regulation and emotion lability/negativity.
Parental Reflective Functioning Questionnaire | Parent is assessed at 3 time-points: pretest (one to two weeks before the first session); posttest (one week after the last session); follow-up (3 months after the last session).
  PRFQ is a questionnaire composed of 18 items that assesses parental reflective functioning in parents. The items are measured on a 7-point Likert scale (1 = strongly disagree; 7 = strongly agree), composed of 3 subscales: pre-mentalizing modes of mental states, certainty about mental states, and interest and curiosity in mental states.
Test of Emotional Comprehension | Child is assessed at 3 time-points: pretest (one to two weeks before the first session); posttest (one week after the last session); follow-up (3 months after the last session).
  TEC is composed of 23 items/stories that asses 9 domains of understanding of emotions in children from 3 to 11 years of age: (1) recognition of emotions based on facial expressions, (2) external causes of emotions, (3) assigning a desire as cause an emotion; (4) the role of believes in determining emotions, (5) the influence of memory in circumstances of assessment of emotional states, (6) the ability to regulate emotions, (7) the ability to hide or conceal an emotion; (8) that a person can have mixed emotions in relation to a given situation, and (9) the role of morality in emotions.

OTHER OUTCOMES:
Sociodemographic Questionnaire | Participants are assessed with the Sociodemographic Questionnaire at 1 time-point: pretest (one to two week before the first session).
  The Sociodemographic Questionnaire was used to collect sociodemographic information of the child and parents - such as gender, age, nationality, household members, socioeconomic level and schooling.
Satisfaction Questionnaire | Participants are assessed with the Satisfaction Questionnaires at 1 time-point: posttest (one week to two after the last session).
  The Satisfaction Questionnaires composed of 14 items each, one for child and another for parent, that seek to assess the level of parental and child satisfaction with MBT-C. 12 Items are scored on a 5-point likert scale (1 = agree completely; 5 = disagree completely) and 2 items are of open response.

CONTACTS AND LOCATIONS:
Overall Officials: Bárbara Figueiredo, PhD, Principal Investigator — Psychology Research Centre (CIPsi), University of Minho
Locations (1):
- University of Minho, Braga, Braga District, Portugal